CLINICAL TRIAL: NCT07316517
Title: Prospective Clinical Study to Evaluate the Safety and Efficacy of Versius in Robot-Assisted Inguinal Hernia Repair Surgery
Brief Title: Versius Clinical Study in Robot Assisted Inguinal Hernia Repair Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CMR Surgical Ltd (Industry)
Collaborators: Division of General Oncologic and Minimally Invasive Surgery, Niguarda Hospital Milan (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA-00615
Record Dates: First submitted 2025-12-05; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Robotic Assisted Inguinal Hernia Repair
Keywords: Versius; Robotic surgery; Inguinal hernia
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surgery with Versius (Experimental)
  Interventions: Device: Versius Surgical System

INTERVENTIONS:
Device: Versius Surgical System — Modular robotic system intended to assist in the accurate control of its surgical endoscopic instruments across a range of surgical procedures.

SUMMARY:
The objective of this clinical trial is to evaluate the safety and efficacy of Versius in Inguinal Hernia repair surgery

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients 22 years of age and older, deemed eligible for elective minimal invasive inguinal Hernia repair surgery.
2. Patients providing written informed consent to participate in the study.

Exclusion Criteria:

1. Patient unwilling to provide informed consent.
2. Medical contraindication for general anaesthesia or minimally invasive procedure.
3. Patient participation in an interventional clinical study that could impact primary outcomes results.
4. Patient who falls into American Society of Anaesthesiologists (ASA) Class IV or above.
5. Patients undergoing a concomitant surgical procedure.
6. Contraindication for undergoing surgery with Versius (bleeding diathesis, active pregnancy or BMI ≥40 kg/m2).

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Success rate | Up to completion of surgery
  Rate of successful completion of robotic assisted surgery as planned without unplanned conversion to other laparoscopic or open surgery
Serious Adverse Event rate | Up to 30 days post procedure
  Rate of total procedure related serious adverse events

SECONDARY OUTCOMES:
Operative time | Up to completion of surgery
  Surgical time from skin incision to skin closure
Estimated blood loss | Up to completion of surgery
  Amount of blood estimated to be lost during surgery (in mL)
Intra-operative adverse events | Up to completion of surgery
  Adverse events that occur during surgery
Blood transfusion | Up to completion of surgery
  Need for blood transfusion during surgery as well as amount transfused
Device deficiencies | Up to completion of surgery
  Any device deficiencies of Versius during surgery
Reoperation within 24 hours | 24 hours post-surgery
  Need for reoperation after initial surgery
Length of hospital stay | Up to post-surgical discharge, i.e. the date when patient is considered sufficiently recovered from surgery to leave hospital, expected to be at most up to 1 month after date of surgery, typically within a few days
  Hospital stay in days from day of surgery until discharge
Adverse events | Up to 30 days post-surgery
  Rate of adverse events
Readmission | Up to 30 days post-surgery
  Hospital readmission after post-surgical discharge
Reoperation within 30 days | Up to 30 days post-surgery
  Need for reoperation as a result of interventional surgery itself or the indication for surgery
Mortality rate | Up to 30 days post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Domenico Antonio Alampi, MD, Principal Investigator — Division of General Oncologic and Minimally Invasive Surgery, Niguarda Hospital Milan
Locations (1):
- Division of General Oncologic and Minimally Invasive Surgery, Niguarda Hospital Milan, Milan, Italy

IPD SHARING:
Plan to Share IPD: No